CLINICAL TRIAL: NCT03499743
Title: Celecoxib Versus Hyoscine Butyl-bromide in Reducing Pain Perception During Copper T380A Intrauterine Device Insertion: a Randomized Double-blind Controlled Trial
Brief Title: Celecoxib Versus Hyoscine Butyl-bromide in Reducing Pain Associated With IUD.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, lecturer in obstetrics and gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IUD insertion pain
Record Dates: First submitted 2018-04-09; First posted 2018-04-17 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: IUD Insertion Pain
MeSH Terms: interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigators who will insert the IUDs and will collect important data, the patients and the statistician who will perform the final data analysis will be blinded to the group allocations
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group1 (hyoscine Butyl-bromide group) (Experimental): group1 will receive hyoscine butyl bromide 10 mg (BUSCOPAN tablets, produced by Chemical Industries Development (CID), Giza - A.R.E. under licence of Boehringer Ingelheim International GmbH - Germany) orally in addition to a placebo similar to Celecoxib 2 hours before IUD insertion.
  Interventions: Drug: hyoscine butyl bromide
- group 3 (PLACEBO GROUP) (Placebo Comparator): will receive a placebo similar to hyoscine butyl bromide in addition to a placebo similar to Celecoxib 2 hours before IUD insertion.
  Interventions: Drug: Placebo Oral Tablet
- group 2(celecoxib group) (Experimental): group 2 will receive Celecoxib 200mg (Celebrex® 200, Pfizer, USA) in addition to a placebo similar to hyoscine butyl bromide 2 hours before IUD insertion.
  Interventions: Drug: Celecoxib 200mg

INTERVENTIONS:
Drug: hyoscine butyl bromide — intake of 10 mg hyoscine butyl bromide (buscopan) orally in addition to a placebo similar to Celecoxib 2 hours before IUD insertion
  Arms: group1 (hyoscine Butyl-bromide group)
Drug: Celecoxib 200mg — Celecoxib 200mg (Celebrex® 200, Pfizer, USA) in addition to a placebo similar to hyoscine butyl bromide
  Arms: group 2(celecoxib group)
Drug: Placebo Oral Tablet — a placebo similar to hyoscine butyl bromide in addition to a placebo similar to Celecoxib.
  Arms: group 3 (PLACEBO GROUP)

SUMMARY:
Many oral analgesic drugs such as the nonsteroidal anti-inflammatory drug (NSAID) are used to relieve pain from gynaecological procedures and dysmenorrhea. Hyoscine-N-butyl bromide, an antispasmodic drug is commonly used for relief of smooth muscle spasms and can be used to alleviate genito-urinary spasm. Some studies reported hyoscine couldn't relieve pain in minor gynaecological procedures. So the efficacy of Hyoscine-N-butyl bromide use is still controversial, and no previous studies investigated its effectiveness for pain relief in IUD insertion procedure.

DETAILED DESCRIPTION:
The study objective is to compare the effectiveness and side effects of oral Celecoxib 200mg versus oral hyoscine butyl bromide 10 mg in reducing pain associated with IUD insertion. the study is an attempt to find the most effective drug with the least possible side effects to be used before IUD insertion.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant nulliparous and parous menstruating women.
* Women who Did not receive any analgesics or misoprostol in the 24 hours prior to insertion.
* Presenting for insertion of CuT380A intrauterine device.
* the absence of contraindication for IUD insertion including positive cultures for gonorrhoea or chlamydia
* the absence of sedative or long-acting narcotics use 48 h before IUD insertion
* No history of severe mental stress in the past two months.

Exclusion Criteria:

* • Allergy to HYOSCINE BUTYLBROMIDE or celecoxib or contraindication to it as paralytic ileus, myasthenia gravis, pyloric stenosis and narrow-angle glaucoma.

  * Women who had been pregnant within the previous four weeks.
  * Women presenting for IUD removal and reinsertion
  * Any uterine abnormalities distorted uterine cavity as congenital anomalies, endometrial lesions, adenomyosis, and submucous myoma.
  * Enrollment in another study.
  * A psychological or neurological disorder associated with altered pain sensation.
  * a history of dysmenorrhea
  * a contraindication for IUD use such as a gynaecological malignancy, pelvic inflammatory disease or undiagnosed abnormal vaginal bleeding.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-05 (Actual)

PRIMARY OUTCOMES:
self-reported pain score | during IUD insertion
  the visual analog scale (VAS ) pain score reported by participants during IUD insertion.Pain scores will be measured using a visual analogue scale (VAS) consisting of a 10 cm horizontal straight line on which 0 cm corresponds to no pain and 10 cm to the worst pain. VAS is rated as 0 for no pain, 1-3 for mild pain, 4-6 for average pain, and 7-9 for severe pain and 10 for extremely severe pain an individual can experience.A research assistant standing beside the woman will hold the VAS sheet for the participant to select the point that corresponds to the level of pain she will experience.

SECONDARY OUTCOMES:
difference in pain score | during tenaculum placement, during sound insertion, and 5 minutes after IUD insertion.
  the pain score at other different points; during tenaculum placement, during sound insertion, and 5 minutes after the end of insertion with a different sheet of paper at every point.
immediate complications related to IUD insertion | 30 minutes after insertion
  the immediate complications related to IUD insertion such as uterine perforation, failure of insertion, vasovagal reaction and bleeding and the number of women who will need analgesics after insertion.

CONTACTS AND LOCATIONS:
Overall Officials: AHMED SAMY, MD, Principal Investigator — Cairo University
Locations (1):
- Obsterics and Gynecology Department, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided